CLINICAL TRIAL: NCT05962671
Title: Opioid-sparing Versus Sevoflurane-based Anesthesia on Early Postoperative Hypoventilation in Patients Undergoing Laparoscopic Bariatric Surgery: Prospective Randomized Study
Brief Title: Opioid-sparing Versus Sevoflurane Anesthesia on Early Postoperative Hypoventilation in Laparoscopic Bariatric Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Samah Mohamed Marie, Doctor resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264MS154/4/23
Record Dates: First submitted 2023-06-24; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia; Hypoventilation; Opioid Use; Bariatric Surgery
MeSH Terms: conditions — Hypoventilation | interventions — Analgesics, Opioid; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-sparing based anesthesia (Active Comparator): Intraoperative opioid-sparing maintenance comprised dexmedetomidine bolus dose of 1 mcg/kg followed by 0.3 mcg/kg/h, propofol 4-8 mg/kg/h and ketamine 25 mg/h for a max of 50 mg during the procedure, targeting bispectral index (BIS) between 45%-60%. The lean body weight will be used for calculation of the drugs.
  Interventions: Drug: Opioid-sparing based anesthesia
- Sevoflurane-based anesthesia (Active Comparator): Intraoperative sevoflurane-based anesthesia, 0.8 to 1.0 Minimum alveolar concentration will be used combined with fentanyl 1 mcg/kg followed by 1 -2 mcg/kg/h and cis-atracurium, to keep bispectral index between 45% to 60%.
  Interventions: Drug: Sevoflurane-based anesthesia

INTERVENTIONS:
Drug: Opioid-sparing based anesthesia — Intraoperative opioid-sparing maintenance comprised dexmedetomidine bolus dose of 1 mcg/kg followed by 0.3 mcg/kg/h, propofol 4-8 mg/kg/h and ketamine 25 mg/h for a max of 50 mg during the procedure, targeting bispectral index (BIS) between 45%-60%. The lean body weight will be used for calculation of the drugs.
  Other Names: Opioid
  Arms: Opioid-sparing based anesthesia
Drug: Sevoflurane-based anesthesia — Intraoperative sevoflurane-based anesthesia, 0.8 to 1.0 Minimum alveolar concentration will be used combined with fentanyl 1 mcg/kg followed by 1 -2 mcg/kg/h and cis-atracurium, to keep bispectral index between 45% to 60%.
  Other Names: Sevoflurane
  Arms: Sevoflurane-based anesthesia

SUMMARY:
Determine the incidence of early post-operative hypoventilation in post-anesthesia care unit (PACU) in patients undergoing laparoscopic bariatric surgery under opioid-sparing compared with sevoflurane-based anesthesia.

DETAILED DESCRIPTION:
The incidence of early postoperative hypoxemia in the literature is diverse, this may be due to multivariable, including patient-related factors, anesthesia-related factors, and surgery-related factors. Because of the controverse regarding the incidence of postoperative hypoxemia and the evidence of anesthetic technique of choice, interest in prevention and early management of early postoperative hypoxemia after laparoscopic bariatric surgery is continued.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients ≥ 18 years
* Admitted to the post anesthesia care unit after bariatric surgery

Exclusion Criteria:

• Preoperative hypoxemia which is determined by a peripheral capillary oxygen saturation (SPO2) reading of < 90% on room air

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Early postoperative hypoventilation | UP to 24 hours Postoperatively
  Early postoperative respiratory hypoventilation will be defined by any of the following parameters:
  Oxygen saturation < 95% for 10 seconds. Respiratory rate < 8 breath/min. Apnea spill > 10 seconds. pain/sedation-mismatch.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: after the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author